CLINICAL TRIAL: NCT02652676
Title: Reversible Pulmonary Artery Banding as Simplified Management of End-stage Dilated Left Ventriculopathy in Early Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5150418
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Acute on Chronic Systolic Congestive Heart Failure
Keywords: Infant Cardiac Transplantation; End-stage Idiopathic Dilated Cardiomyopathy; Mechanical Circulatory Device; End Stage Dilated Left Ventriculopathy; Acute-on-Chronic Left Ventricular Failure
MeSH Terms: interventions — Biocompatible Materials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reversible Pulmonary Artery Banding Procedure (Experimental): The addition of afterload Reversible Pulmonary Artery Banding to a normal-functioning right ventricle (in the setting of end-stage dilated cardiomyopathy) shifts the inter-ventricular septum toward the midline, thus significantly improving left ventricular geometry and function. It permits the infant or young child to operate from a much improved position on Starling's curve with gradual resolution of congestive heart failure and the potential for lethal ventricular dysrhythmia. An abundance of progenitor myocytes known to exist within the myocardium of this patient age group may then contribute to "permanent" left ventricular restoration.
  Interventions: Procedure: Reversible Pulmonary Artery Banding; Procedure: GORE-TEX DualMesh EMERGE PLUS Biomaterial

INTERVENTIONS:
Procedure: Reversible Pulmonary Artery Banding — A sternotomy incision is used for application of the rPAB. Tightening is under echocardiographic control until the inter-ventricular septum becomes a midline structure. Myocardial function is augmented with inotropic and vasodilator agents that are weaned after 2-4 weeks. The infant is separated from mechanical ventilation within the first week, and enteric feeding is resumed. The infant is discharged on oral medications, with follow-ups. Band enlargement is in stages as a balloon catheter-based procedure if a finding of increasing right ventricular dilation, onset or worsening tricuspid valve regurgitation, or a gradual late increase in plasma B-type natriuretic peptide (BNP) levels, opting for a mild residual right ventricle-main pulmonary artery pressure gradient of 15-30 mmHg.
  Other Names: rPAB
Procedure: GORE-TEX DualMesh EMERGE PLUS Biomaterial — The study is being conducted to evaluate the procedure, not the materials being used. The study uses the patch as materials to create the band around the pulmonary artery which is currently done routinely off label. The patch is approved as a cardiovascular patch. FDA 501(k) K032168.
  Other Names: Gortex Cardiovascular Patch

SUMMARY:
The purpose of this study is to: 1) Remodel and restore left ventricular geometry and function. 2) Avoid the need for mechanical circulatory support (MCS) and/or cardiac transplantation (CT). 3) Confirm the outcomes of a pilot study completed in Germany and reported in The Journal of Heart and Lung Transplantation in May 2013.

DETAILED DESCRIPTION:
The study infant will undergo cardiac catheterization and myocardial biopsy before pulmonary artery banding and at appropriate intervals during follow-up surveillance by the interventional cardiologist. Patients will be "listed" for heart transplantation, and rPAB will be applied in lieu of mechanical circulatory support or as an alternative to already existing mechanical circulatory support, in the form of extracorporeal mechanical oxygen (ECMO). Myocardial biopsies will be flash frozen for storage and eventual probing for cell type (mature or stem) as part of a separate study.

The addition of afterload rPAB to a normal-functioning right ventricle (in the setting of end-stage dilated cardiomyopathy) shifts the inter-ventricular septum toward the midline, thus significantly improving left ventricular geometry and function. It permits the infant or young child to operate from a much improved position on Starling's curve with gradual resolution of congestive heart failure and the potential for lethal ventricular dysrhythmia. An abundance of progenitor myocytes known to exist within the myocardium of this patient age group may then contribute to "permanent" left ventricular restoration.

A sternotomy incision is used for application of the rPAB. The band is tightened under echocardiographic control until the inter-ventricular septum becomes a midline structure. Myocardial function is augmented with inotropic and vasodilator agents. These agents are weaned off gradually over a period of 2-4 weeks. The infant is separated from mechanical ventilation within the first post-rPAB week, and enteric feeding is resumed. The infant is discharged on oral medications, and is kept under frequent clinical surveillance.

As the infant grows, the rPAB becomes relatively more obstructive to right ventricular outflow. Based on a finding of increasing right ventricular dilation, onset or worsening tricuspid valve regurgitation, or a gradual late increase in plasma B-type natriuretic peptide (BNP) levels, the band may be loosened in stages as a balloon catheter-based procedure. Band enlargement may be accomplished in stages, ultimately opting for a mild residual right ventricle-main pulmonary artery pressure gradient of 15-30 mmHg.

The infants' short- and long-term surveillance will include clinical examination, height, weight, cardiac catheterization, electrocardiogram, echocardiogram, chest x-ray, and plasma BNP levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-4 years
2. Isolated, idiopathic left-ventricular end-stage dilated cardiomyopathy or a Left Ventricular End-Diastolic Diameter (LVEDD) Z-score > 4.5; Ejection Fraction (EF) < 30%
3. Acceptable candidate for mechanical circulatory support and/or cardiac transplantation
4. Preserved right-ventricular function
5. Clinical functional status IV (hospitalized)
6. Parental consent

Exclusion Criteria:

1. Biventricular end-stage dilated cardiomyopathy
2. Proven or suspected myocarditis
3. Concomitant structural (congenital) heart disease
4. Moderate-severe tricuspid valve regurgitation
5. Pulmonary hypertension out of proportion with left-ventricular end-stage cardiomyopathy
6. Hereditary disease associated with bi-ventricular dysfunction
7. Age greater than 4 years
8. No parental consent

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Surgical Success | 5 years
  positive surgical outcome, the survival of the patient, the lack of a need for mechanical circulatory support or heart transplant, and improved left ventricular function

SECONDARY OUTCOMES:
All Cause Mortality | 5 years
  Total number of deaths due to non-cardiac open vs minimally invasive thoracic surgery.
Persistent Heart Failure | 5 years
  Described as having an NYHA of greater than II.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Martens, MD, PhD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States

REFERENCES:
- [Background] Arbustini E, Weidemann F, Hall JL. Left ventricular noncompaction: a distinct cardiomyopathy or a trait shared by different cardiac diseases? J Am Coll Cardiol. 2014 Oct 28;64(17):1840-50. doi: 10.1016/j.jacc.2014.08.030. Epub 2014 Oct 21. PMID 25443708
- [Background] Bailey LL. Back to the future! Bold new indication for pulmonary artery banding. J Heart Lung Transplant. 2013 May;32(5):482-3. doi: 10.1016/j.healun.2013.03.001. No abstract available. PMID 23570740
- [Background] Brancaccio G, Amodeo A, Ricci Z, Morelli S, Gagliardi MG, Iacobelli R, Michielon G, Picardo S, Parisi F, Pongiglione G, Di Donato RM. Mechanical assist device as a bridge to heart transplantation in children less than 10 kilograms. Ann Thorac Surg. 2010 Jul;90(1):58-62. doi: 10.1016/j.athoracsur.2010.03.056. PMID 20609748
- [Background] Everett BM, Berger JS, Manson JE, Ridker PM, Cook NR. B-type natriuretic peptides improve cardiovascular disease risk prediction in a cohort of women. J Am Coll Cardiol. 2014 Oct 28;64(17):1789-97. doi: 10.1016/j.jacc.2014.04.089. Epub 2014 Oct 21. PMID 25443700
- [Background] Julious SA. Two-sided confidence intervals for the single proportion: comparison of seven methods by Robert G. Newcombe, Statistics in Medicine 1998; 17:857-872. Stat Med. 2005 Nov 15;24(21):3383-4. doi: 10.1002/sim.2164. No abstract available. PMID 16206245
- [Background] Miyamoto SD, Karimpour-Fard A, Peterson V, Auerbach SR, Stenmark KR, Stauffer BL, Sucharov CC. Circulating microRNA as a biomarker for recovery in pediatric dilated cardiomyopathy. J Heart Lung Transplant. 2015 May;34(5):724-33. doi: 10.1016/j.healun.2015.01.979. Epub 2015 Jan 30. PMID 25840506
- [Background] Ross RD. The Ross classification for heart failure in children after 25 years: a review and an age-stratified revision. Pediatr Cardiol. 2012 Dec;33(8):1295-300. doi: 10.1007/s00246-012-0306-8. Epub 2012 Apr 5. PMID 22476605
- [Background] Schranz D, Veldman A, Bartram U, Michel-Behnke I, Bauer J, Akinturk H. Pulmonary artery banding for idiopathic dilative cardiomyopathy: a novel therapeutic strategy using an old surgical procedure. J Thorac Cardiovasc Surg. 2007 Sep;134(3):796-7. doi: 10.1016/j.jtcvs.2007.04.044. No abstract available. PMID 17723838
- [Background] Schranz D, Rupp S, Muller M, Schmidt D, Bauer A, Valeske K, Michel-Behnke I, Jux C, Apitz C, Thul J, Hsu D, Akinturk H. Pulmonary artery banding in infants and young children with left ventricular dilated cardiomyopathy: a novel therapeutic strategy before heart transplantation. J Heart Lung Transplant. 2013 May;32(5):475-81. doi: 10.1016/j.healun.2013.01.988. Epub 2013 Feb 12. PMID 23410738